CLINICAL TRIAL: NCT03422276
Title: Improving Transition From Acute to Post-Acute Care Following Traumatic Brain Injury
Brief Title: Brain Injury Rehabilitation Improving the Transition Experience
Acronym: BRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Moss Rehabilitation Research Institute (Other); Ohio State University (Other); Baylor Institute for Rehabilitation (Other); Indiana University School of Medicine (Other); Craig Hospital (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor, School of Medicine: Rehabilitation Medicine:Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00002859; PCS-1604-35115 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: Transition; Rehabilitation Discharge
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study uses masked outcome assessment, which means study researchers will make every effort to ensure that staff members who collect outcomes data from both patient and caregiver participants at 3-, 6-, 9- and 12 months are unaware of patient participants' treatment group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Discharge Plan (Active Comparator): Commission on Accreditation of Rehabilitation Facilities (CARF) standards for discharge following an inpatient rehabilitation stay for a traumatic brain injury, including patient and family education, written discharge care instructions, and telephone follow up from a clinical provider.
  Interventions: Other: Rehabilitation Discharge Plan
- Rehabilitation Transition Plan (Active Comparator): Approximately 12 scheduled contacts from a TBI care manager 6 months following discharge in addition to the CARF standards for discharge.
  Interventions: Other: Rehabilitation Transition Plan

INTERVENTIONS:
Other: Rehabilitation Discharge Plan — CARF standards for discharge following an inpatient rehabilitation stay for a traumatic brain injury. This approach may include the following:
  1. patient and family education about TBI, both general and individualized to each person's symptoms and level of function, as well as education on medications and symptoms to monitor following discharge;
  2. written discharge care instructions, including recommended appointments with primary care, rehabilitation medicine and outpatient therapies, and medication list which are reviewed with the patient and family prior to discharge; and
  3. a phone call from an inpatient care provider within a few days of discharge to address any immediate problems and ensure that equipment has arrived, medications are being taken, etc.
  Arms: Rehabilitation Discharge Plan
Other: Rehabilitation Transition Plan — Participants and their caregivers (if applicable) randomized to the Rehabilitation Transition Plan group will receive up to 12 scheduled contacts 6 months post-discharge from a TBI care manager familiar with the care and resource networks at the respective sites. The contacts will at minimum be by telephone, although a HIPAA-compliant video conferencing option will also be available.
  The content of these contacts will include:
  1. Particularly in the first few calls, review of discharge plans and assistance and/or directive problem-solving around any obstacles to following discharge plans;
  2. Assessment of unmet needs, developed into a standard checklist of areas of need that are relevant to TBI, culled from literature on need fulfillment in this population.
  Arms: Rehabilitation Transition Plan

SUMMARY:
Each year, about 2.8 million people sustain a traumatic brain injury (TBI) in the United States, and at least 25 percent of these injuries are classified as moderate to severe. Nearly half of those hospitalized for TBI have long-term disability. Most have psychological, physical, social, or work-related problems, which often become chronic. By talking with patients and family members, we found that returning to daily activities and regaining quality of life are major concerns. Outcomes are affected by the type and severity of the TBI, but the type of treatment someone with TBI receives is also important. What resources are available, whether providers are experienced with the problems associated with TBI, and how much treatment is available can affect outcomes as well.

Currently, inpatient rehabilitation professionals are told to give people with TBI information, reassurance, advice, and referral resources. Some promising ways of helping people with TBI include using telephone and other mobile devices to reach patients after they leave the hospital, to regularly assess their individual needs and help them coordinate their health care, and to provide the information and resources that they need. These new strategies may lead to earlier return to activities and improved quality of life. No studies have compared the standard approach to discharge care with an approach that uses telecare to provide information and care coordination after discharge from inpatient rehabilitation for TBI.

The main goal of this project is to find out how improving the transition from the hospital to outpatient care can improve the lives of people with moderate to severe TBI and achieve better results that are important to patients with TBI, their families, and healthcare providers. In this study, patients with TBI who are discharged from inpatient rehabilitation at one of six national TBI Model Systems sites (University of Washington, Indiana University, Ohio State University, Mount Sinai Hospital, Moss Rehabilitation, and Baylor Institute for Rehabilitation) will be randomized (like the flip of a coin) to either the standard discharge plan or the standard discharge plan with additional telephone follow up from a TBI care manager for the first 6 months after discharge. The project team will compare patient and caregiver functioning and quality of life at 3, 6, 9, and 12 months after hospital discharge in these two groups.

DETAILED DESCRIPTION:
Screening

The screening process involves a review of medical records by our research staff for patients with a diagnosis of TBI, or suspected TBI, (see inclusion/exclusion for further detail) who are admitted to the inpatient rehabilitation unit at the study sites.

Recruitment

Patient Participants: If a potential participant meets eligibility criteria based on medical record review, research staff will approach him/her on the inpatient rehabilitation unit to determine whether the patient is cognitively capable of providing consent by administering a measure of orientation/ emergence from PTA. If the patient is deemed oriented, the research staff will introduce the study using a talking points script, and if the potential participant is interested, provide him/her with a brochure and a consent form.

Research staff will initiate the informed consent process if: a) the patient is deemed oriented per definition above, and b) the patient expresses interest in participating. Research staff will visit the patient on a subsequent day and re-administer the orientation test prior to consent if needed.

If the patient is not deemed oriented as per the outline above, the patient is deemed not yet oriented and unable at that time to provide informed consent. Research staff may administer the orientation test multiple times to determine capacity to consent. Research staff may talk with a Legally Authorized Representative (LAR) if one is willing and available to attempt to obtain their consent if a patient is not deemed oriented prior to discharge.

The investigators plan to enroll a total of 900 patient participants.

Caregiver Participants:

Caregiver participants will be those individuals who will have primary care giving responsibility following rehabilitation care discharge of patients with moderate to severe TBI. Caregivers may be recruited while the patient is in the hospital or by telephone, if not available during hospitalization. Research staff may enroll more than one individual as a caregiver following subject enrollment should a different individual assume the role of caregiver at a later time point.

The investigators plan to enroll a total of 607 caregiver participants.

Basic Demographic Information: All Potential Patient Participants

Basic demographic information including age, sex, and race will be collected via medical record review without consent from all patients including those who do not enroll to determine differences between enrolled patients participants and those who do not enroll.

Consent

For patient participants, the informed consent process will take place during the participants inpatient rehabilitation stay with our research staff while they are inpatients.

Potential participants will be fully informed of all risks and benefits prior to giving their written informed consent and prior to enrollment in the study. Participants may take time to think about participating and render a decision in a subsequent visit. Potential participants will be asked to repeat back understanding of this material as necessary.

Research staff will also review a HIPAA authorization form with the participant that permits research staff to collect data from his/her medical records regarding injury and medical history.

Caregiver Participants: Caregiver participants may be initially recruited by telephone or in person. Caregivers will provide written consent if enrolled in person.

All participants approached for possible enrollment in this study will be clearly informed that if they choose not to participate in this project, they and/or their loved one will still be able to receive any of the routine medical and rehabilitation services available to them. They will be informed that their participation is voluntary and that they may withdraw their consent and discontinue participation in the study at any time. Any new information developed during the course of the study that might affect a participant's understanding of the research and willingness to continue to participate will be brought to their attention by study staff.

Baseline Assessment

Contact Information Sheet Research staff will collect the following information from both caregiver and patient participants: (1) contact information; (2) best way to reach an individual if they have more than one line; best times/days to reach participant; and (3) names and contact information of people staff are allowed to contact if participant is lost to follow-up or otherwise cannot be contacted (i.e. collateral contacts).

Baseline Information: Demographic and injury related data will be collected from the electronic medical record, and additional demographic and clinical history will be collected in interview format. A cognitive assessment focused on memory, concentration, and problem solving will be given. These data will be entered in de-identified form into the NDSC centralized database by research staff.

Discharge Information: Research staff will collect information from a patient participant's medical record regarding the presence/absence of recommended and/or scheduled appointments to different medical disciplines/services. Specific information regarding the recommended/scheduled appointments (e.g. name, phone number, email address, date of scheduled appointment, etc.) of patient participants randomized to the rehabilitation transition phase (RTP) group will be stored locally in a database used by the TBI care managers for referential purposes.

The investigators will collect information regarding the nature of the caregiver's relationship to the patient participant, as well as basic demographic information. These data will be entered in de-identified form into the NDSC centralized database by research staff.

Randomization/ Post-Discharge Transition Phase

After the patient participant has been discharged, s/he will be randomly assigned 1:1 into one of two study arms: Rehabilitation Discharge Plan (RDP) group or the Rehabilitation Transition Plan (RTP) group.

The investigators will stratify randomization on study site and discharge destination (another facility vs. home/ community). Once randomization occurs, their random assignment will be communicated to the TBI Care Manager (TCM). The TCM will then send out a letter to the patient participant and caregiver (if applicable).

RTP Process Variables

Individual elements of the RTP will be measured as they are administered to each patient/ caregiver or other recipient in the form of a treatment note as captured in a secure database, incorporating documentation elements used in the field. Measures will include the clock time devoted to each contact, the recipient of each contact, total number of attempts/contacts, the type of need or issue discussed, and actions planned and implemented.

Follow Up Data Collection

3, 6, 9 and 12 Months Post Hospital Discharge: Patient Participant The 3, 6, 9 and 12 month post-hospital discharge questionnaire will take approximately 45-60 minutes to complete, and will be completed by phone or in person. This questionnaire includes both the primary and secondary outcomes described below.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a moderate-to-severe TBI defined by TBIMS and this study as damage to brain tissue caused by an external mechanical force as evidenced by medically documented loss of consciousness or post-traumatic amnesia (PTA) due to brain trauma or by objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination. Potential participants must meet at least one of the following criteria to be considered experiencing a moderate-to-severe TBI:

   1. PTA>24 hours;
   2. Trauma related intracranial neuroimaging abnormalities;
   3. Loss of consciousness exceeding 30 minutes (unless due to sedation or intoxication); or
   4. Glasgow Coma Scale in the emergency department of less than 13 (unless due to intubation, sedation, or intoxication).
2. English speaking (we will track non-enrollment due to other language to determine common languages and have consumer dissemination materials translated for more broad use if time and resources permit.);
3. At least 18 years old;
4. Will be discharged from inpatient rehabilitation to community (private residence, adult home, hotel, homeless) or facility (nursing home, subacute care i.e. skilled nursing facility);
5. Current admission to inpatient rehabilitation considered their first comprehensive rehabilitation experience, or extension thereof for most recent TBI (e.g. admitted to inpatient rehabilitation, discharged to acute care, then returns to inpatient rehabilitation to complete their initial stay);
6. Able to provide informed consent, or if unable to provide consent have family or legal guardian to provide informed consent for the patient.

Inclusion Criteria- Caregiver Participants:

1. Individuals who will have primary care giving responsibility post rehabilitation care discharge of enrolled patient participants;
2. English speaking (we will track non-enrollment due to other language to determine common languages and have consumer dissemination materials translated for more broad use if time and resources permit.);
3. At least 18 years old;
4. Able to provide informed consent.

Exclusion Criteria:

Exclusion criteria- Patient Participants:

1. We will not enroll individuals who are in law enforcement custody at admission to the designated rehabilitation unit or who are taken into custody prior to discharge from the designated rehabilitation unit due to federal restrictions on inclusion of prisoners in research.
2. We will not enroll individuals who do not have access to a phone.
3. We will not enroll individuals who are unable to complete study procedures due to cognitive/verbal limitations AND do not have a proxy to assist with study procedures.

Exclusion criteria- Caregiver Participants:

1. We will not enroll individuals who are in law enforcement custody due to federal restrictions on inclusion of prisoners in research.
2. We will not enroll individuals who do not have access to a phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1555 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Hoffman, PhD, Principal Investigator — University of Washington; Jesse Fann, MD, MPH, Principal Investigator — University of Washington
Locations (6):
- United States (6):
  - Indiana University School of Medicine/ Rehabilitation Hospital of Indiana, Indianapolis, Indiana
  - Mount Sinai Health System (NY), New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Moss Rehab Hospital, Elkins Park, Pennsylvania
  - Baylor Institute for Rehabilitation, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Fann JR, Hart T, Ciol MA, Moore M, Bogner J, Corrigan JD, Dams-O'Connor K, Driver S, Dubiel R, Hammond FM, Kajankova M, Watanabe TK, Hoffman JM. Improving transition from inpatient rehabilitation following traumatic brain injury: Protocol for the BRITE pragmatic comparative effectiveness trial. Contemp Clin Trials. 2021 May;104:106332. doi: 10.1016/j.cct.2021.106332. Epub 2021 Feb 27. PMID 33652127
- [Derived] Moore M, Kempthorne L, Fann JR, Shulein O, Dams-O'Connor K, Kajankova M, Conrick KM, Seeliger J, Hoffman JM. Patient and Caregiver Satisfaction With the Brain Injury Rehabilitation: Improving the Transition Experience (BRITE) Intervention. J Head Trauma Rehabil. 2024 Nov-Dec 01;39(6):E550-E563. doi: 10.1097/HTR.0000000000000949. Epub 2024 May 13. PMID 38758094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient participants were recruited from 6 IPR facilities starting in Feb 2018 through Aug 2021. Caregivers (CG) of enrolled patients were recruited from the first patient enrollment through the end of patient participation. The final CG enrolled in February 2022. Patients could have more than one CG enrolled in the study due to changes in primary caregiver responsibility. Only one CG completed each follow up (max N at any follow up 591), but a total of 611 CG were enrolled throughout the study.
Pre-assignment Details: 11 patients were enrolled but not randomized in the study for the following reasons: Determined to be ineligible, death, withdrew, and other. The majority (8) were determined to be ineligible. 8 caregivers were enrolled to patients that were not randomized. So a total of 19 of the 1555 enrolled patients and caregivers were not part of the randomized cohort.
Groups:
- Rehabilitation Discharge Plan: Commission on Accreditation of Rehabilitation Facilities (CARF) standards for discharge following an inpatient rehabilitation stay for a traumatic brain injury, including patient and family education, written discharge care instructions, and telephone follow up from a clinical provider.
  Rehabilitation Discharge Plan: CARF standards for discharge following an inpatient rehabilitation stay for a traumatic brain injury. This approach may include the following:
  1. patient and family education about TBI, both general and individualized to each person's symptoms and level of function, as well as education on medications and symptoms to monitor following discharge;
  2. written discharge care instructions, including recommended appointments with primary care, rehabilitation medicine and outpatient therapies, and medication list which are reviewed with the patient and family prior to discharge; and
  3. a phone call from an inpatient care provider within a few days of discharge to address any immediate problems and ensure that equipment has arrived, medications are being taken, etc.
- Rehabilitation Transition Plan: Approximately 12 scheduled contacts from a TBI care manager 6 months following discharge in addition to the CARF standards for discharge.
  Rehabilitation Transition Plan: Participants and their caregivers (if applicable) randomized to the Rehabilitation Transition Plan group will receive up to 12 scheduled contacts 6 months post-discharge from a TBI care manager familiar with the care and resource networks at the respective sites. The contacts will at minimum be by telephone, although a HIPAA-compliant video conferencing option will also be available.
  The content of these contacts will include:
  1. Particularly in the first few calls, review of discharge plans and assistance and/or directive problem-solving around any obstacles to following discharge plans;
  2. Assessment of unmet needs, developed into a standard checklist of areas of need that are relevant to TBI, culled from literature on need fulfillment in this population.
- Rehabilitation Discharge Plan - Caregivers: Caregivers of patients randomized to the Rehabilitation Discharge Plan (RDP) group
- Rehabilitation Transition Plan - Caregivers: Caregivers of patients randomized to the Rehabilitation Transition Plan (RTP) group
Period: Overall Study
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Started | 462 | 463 | 296 (For 13 of the 296, two different people were enrolled as caregiver at different points in the patient's study participation but a max of 296 could complete data at any time point.) | 295 (For 7 of the 295, two different people were enrolled as caregiver at different points in the patient's study participation but a max of 295 were available to complete at any given time point.)
Completed | 407 | 405 | 246 | 254
Not Completed | 55 | 58 | 50 | 41
Not completed — Withdrawal by Subject | 21 | 25 | 14 | 16
Not completed — Death | 14 | 21 | 3 | 1
Not completed — Discontinued, ineligible | 4 | 3 | 0 | 0
Not completed — Lost to Follow-up | 15 | 8 | 13 | 4
Not completed — Discontinued, researcher decided not in participant's best interest | 1 | 0 | 1 | 0
Not completed — Incarcerated prior to first follow-up | 0 | 1 | 0 | 0
Not completed — Discontinued, no longer caregiver for patient participant | 0 | 0 | 10 | 3
Not completed — Discontinued, for caregiver, death of patient participant | 0 | 0 | 8 | 17
Not completed — Discontinued, for caregiver, patient participant was determined to be ineligible | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There are 20 additional caregiver participants that were enrolled to patient participants who already had one caregiver enrolled. 13 additional caregivers were enrolled to patient participants in RDP and 7 in RTP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers | Total
Number analyzed (Participants) | 462 | 463 | 309 | 302 | 1536
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Patient and Caregiver participants were analyzed separately, so each group is presented in a separate row.
  years
    Patients: number analyzed (Participants) | 462 | 463 | 0 | 0 | 925
    Patients | 48 (20) | 47 (20) |  |  | 47 (20)
    Caregivers: number analyzed (Participants) | 0 | 0 | 309 | 302 | 611
    Caregivers |  |  | 50 (15) | 51 (13) | 51 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 114 | 218 | 225 | 691
  Male | 328 | 349 | 91 | 77 | 845
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Difference for RDP and RTP is due to missing values. For RDP-Caregivers and RTP-Caregivers, this item was not collected.
  Participants
    number analyzed (Participants) | 449 | 452 | 0 | 0 | 901
    Hispanic or Latino | 47 | 29 |  |  | 76
    Not Hispanic or Latino | 402 | 423 |  |  | 825
    Unknown or Not Reported | 0 | 0 |  |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Difference is due to missing values in measure.
  Participants
    Race: number analyzed (Participants) | 458 | 457 | 303 | 295 | 1513
    Race: White | 296 | 314 | 221 | 214 | 1045
    Race: Black | 81 | 79 | 42 | 44 | 246
    Race: Hispanic | 53 | 33 | 24 | 13 | 123
    Race: Other | 28 | 31 | 16 | 24 | 99
Region of Enrollment [Number; unit: participants]
  United States | 462 | 463 | 309 | 302 | 1536
Education Level [Count of Participants; unit: Participants] — Population: Differences are due to missing values.
  Participants
    number analyzed (Participants) | 454 | 457 | 300 | 293 | 1504
    Less than High School | 66 | 59 | 13 | 11 | 149
    HS Diploma or GED | 161 | 152 | 85 | 79 | 477
    Some College | 126 | 118 | 93 | 84 | 421
    College or more | 101 | 128 | 109 | 119 | 457
Married/Partner, yes [Count of Participants; unit: Participants] — Population: Differences are due to missing values.
  Participants
    number analyzed (Participants) | 458 | 458 | 303 | 296 | 1515
    (all) | 159 | 189 | 193 | 194 | 735
Competitively employed, yes [Count of Participants; unit: Participants] — Population: Differences are due to missing values.
  Participants
    number analyzed (Participants) | 456 | 458 | 302 | 296 | 1512
    (all) | 268 | 284 | 202 | 203 | 957
Earnings [Count of Participants; unit: Participants] — Population: Differences are due to missing values. Caregivers that had no annual earnings are included in the missing values.
  Participants
    number analyzed (Participants) | 418 | 414 | 201 | 209 | 1242
    None | 167 | 155 | 0 | 0 | 322
    Less than 30k | 84 | 84 | 41 | 54 | 263
    30K to less than 60K | 87 | 89 | 84 | 70 | 330
    60K or more | 80 | 86 | 76 | 85 | 327
English spoken at home, yes [Count of Participants; unit: Participants] — Population: Differences for RDP and RTP are due to missing values. Caregiver data was not collected for this measure.
  Participants
    number analyzed (Participants) | 459 | 458 | 0 | 0 | 917
    (all) | 433 | 428 |  |  | 861
Residence zone of discharge [Count of Participants; unit: Participants] — Population: Differences for RDP and RTP are due to missing values. Caregiver data was not collected for this measure.
  Participants
    number analyzed (Participants) | 453 | 453 | 0 | 0 | 906
    Urban/Suburban | 314 | 301 |  |  | 615
    Rural | 139 | 152 |  |  | 291
Ever used illicit drugs, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 452 | 454 | 0 | 0 | 906
    (all) | 102 | 120 |  |  | 222
Ever had psychiatric hospitalization, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers
  Participants
    number analyzed (Participants) | 456 | 457 | 0 | 0 | 913
    (all) | 39 | 40 |  |  | 79
Ever had mental health treatment, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 456 | 457 | 0 | 0 | 913
    (all) | 112 | 136 |  |  | 248
Ever attempted suicide, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 452 | 456 | 0 | 0 | 908
    (all) | 25 | 35 |  |  | 60
Ever served in military, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 457 | 458 | 0 | 0 | 915
    (all) | 55 | 60 |  |  | 115
Living alone at discharge, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 459 | 459 | 0 | 0 | 918
    (all) | 23 | 15 |  |  | 38
Discharge to facility, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  Participants
    number analyzed (Participants) | 462 | 463 | 0 | 0 | 925
    (all) | 89 | 89 |  |  | 178
Spinal Cord Injury (SCI), yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 459 | 457 | 0 | 0 | 916
    (all) | 58 | 58 |  |  | 116
Limitations prior to injury, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  Participants
    number analyzed (Participants) | 457 | 458 | 0 | 0 | 915
    (all) | 222 | 209 |  |  | 431
Alcohol use problem [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not collected from caregivers.
  Participants
    number analyzed (Participants) | 428 | 437 | 0 | 0 | 865
    (all) | 111 | 97 |  |  | 208
Cause of injury [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  Participants
    number analyzed (Participants) | 456 | 457 | 0 | 0 | 913
    Vehicle (includes pedestrian/bike) | 232 | 248 |  |  | 480
    Fall | 168 | 146 |  |  | 314
    Violence | 40 | 41 |  |  | 81
    Other | 16 | 22 |  |  | 38
Rehab length of stay [Mean (Standard Deviation); unit: days] — Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  days
    number analyzed (Participants) | 459 | 459 | 0 | 0 | 918
    (all) | 26 (23) | 26 (26) |  |  | 26 (24)
Functional Independence Measure (FIM) Cognitive subscale at discharge [Mean (Standard Deviation); unit: units on a scale] — The Functional Independence Measure (FIM) is an instrument that measures level of disability and required assistance. It is an 18-item scale with motor and cognitive subscales. This captures the cognitive subscale score at discharge (the baseline time point), which can range from 5-35. Higher scores indicate higher functional independence. Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  units on a scale
    number analyzed (Participants) | 419 | 420 | 0 | 0 | 839
    (all) | 23 (6.7) | 22.9 (6.7) |  |  | 23 (6.7)
Functional Independence Measure (FIM) Motor subscale at discharge [Mean (Standard Deviation); unit: units on a scale] — The Functional Independence Measure (FIM) is an instrument that measures level of disability and required assistance. It is an 18-item scale with motor and cognitive subscales. This captures the motor subscale score at discharge (the baseline time point), which can range from 13-91. Higher scores indicate higher functional independence. FIM Motor was either collected with FIM instrument or was transformed from the Continuity Assessment Record and Evaluation (CARE) tool to FIM Motor, according to the crosswalk developed by Dave Mellick. Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  units on a scale
    number analyzed (Participants) | 455 | 455 | 0 | 0 | 910
    (all) | 63.3 (20) | 64.1 (19.7) |  |  | 63.7 (19.8)
Insurance type, yes [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  Participants
    number analyzed (Participants) | 459 | 459 | 0 | 0 | 918
    Medicare | 118 | 98 |  |  | 216
    Medicaid | 108 | 118 |  |  | 226
    Private/self | 180 | 199 |  |  | 379
    Other, Workers Comp, Charity | 53 | 44 |  |  | 97
Glasgow Coma Scale (GCS) Severity Score [Count of Participants; unit: Participants] — Population: Differences for RDP and RTP are due to missing values. For RDP - Caregivers and RTP - Caregivers, this measure is not applicable.
  Participants
    number analyzed (Participants) | 427 | 416 | 0 | 0 | 843
    Severe (3-8) | 55 | 65 |  |  | 120
    Moderate (9-12) | 41 | 42 |  |  | 83
    Mild (13-15) | 159 | 127 |  |  | 286
    Sedated/Intubated | 172 | 182 |  |  | 354
Severity according to time in PTA [Count of Participants; unit: Participants] — Population: Differences in RDP and RTP are due to missing values. Not applicable to caregivers.
  Participants
    number analyzed (Participants) | 420 | 416 | 0 | 0 | 836
    0 to 24h (mild) | 73 | 70 |  |  | 143
    25h to 7 days (moderate) | 43 | 47 |  |  | 90
    More than 7 days (severe) | 304 | 299 |  |  | 603
Country of birth, USA [Count of Participants; unit: Participants] — Population: Patient data was not collected for this measure. Differences for caregiver groups are due to missing values.
  Participants
    number analyzed (Participants) | 0 | 0 | 304 | 295 | 599
    (all) |  |  | 278 | 260 | 538
Relationship to patient [Count of Participants; unit: Participants] — Population: Patient data was not collected for this measure. Measure only included in/or applicable to caregiver demographics. Differences for caregiver groups are due to missing values.
  Participants
    number analyzed (Participants) | 0 | 0 | 304 | 295 | 599
    Spouse |  |  | 117 | 114 | 231
    Parent |  |  | 86 | 89 | 175
    Daughter or Son |  |  | 48 | 32 | 80
    Boyfriend, Girlfriend, Fiancé, Partner |  |  | 23 | 20 | 43
    Sibling |  |  | 19 | 23 | 42
    Other relative |  |  | 7 | 9 | 16
    Friend |  |  | 1 | 4 | 5
    Other |  |  | 3 | 4 | 7
Living in same household, yes [Count of Participants; unit: Participants] — Population: Patient data was not collected for this measure. Measure only included in/or applicable to caregiver demographics. Differences for caregiver groups are due to missing values.
  Participants
    number analyzed (Participants) | 0 | 0 | 303 | 295 | 598
    (all) |  |  | 195 | 189 | 384
Living in private residence, yes [Count of Participants; unit: Participants] — Population: Patient data was not collected for this measure. Measure only included in/or applicable to caregiver demographics. Differences for caregiver groups are due to missing values.
  Participants
    number analyzed (Participants) | 0 | 0 | 303 | 295 | 598
    (all) |  |  | 302 | 294 | 596
Person living with caregiver [Count of Participants; unit: Participants] — Population: Patient data was not collected for this measure. Measure only included in/or applicable to caregiver demographics. Differences for caregiver groups are due to missing values.
  Participants
    number analyzed (Participants) | 0 | 0 | 303 | 295 | 598
    Spouse |  |  | 188 | 191 | 379
    Significant Other |  |  | 32 | 27 | 59
    Alone |  |  | 23 | 24 | 47
    Child/Children |  |  | 15 | 27 | 42
    Other relative(s)/Adult Children |  |  | 23 | 13 | 36
    Parent(s) |  |  | 16 | 11 | 27
    Siblings |  |  | 3 | 2 | 5
    Roommate(s) or Friend(s) |  |  | 3 | 0 | 3
Years (decimal) know the patient [Mean (Standard Deviation); unit: years] — Population: Patient data was not collected for this measure. Measure only included in/or applicable to caregiver demographics. Differences for caregiver groups are due to missing values.
  years
    number analyzed (Participants) | 0 | 0 | 301 | 289 | 590
    (all) |  |  | 30.1 (15.6) | 30.0 (15.6) | 30.1 (15.6)
Years (decimal) lived in the same house [Mean (Standard Deviation); unit: years] — Population: Patient data was not collected for this measure. Measure only included in/or applicable to caregiver demographics. Differences for caregiver groups are due to removing those that did not live in the same household and missing values.
  years
    number analyzed (Participants) | 0 | 0 | 207 | 203 | 410
    (all) |  |  | 19.3 (16.3) | 18.4 (14.6) | 18.8 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Participation Assessment With Recombined Tools - Objective 17 (PART-O-17)
Description: The Participation Assessment with Recombined Tools - Objective 17 (PART-O-17) assesses participation in usual roles and social activities. There are 17 items with 0-5 response scales. Those items are combined and averaged into three domain subscale scores that range from 0-5: Productivity (3 items), Social Relations (7 items), and Out and About (7 items). The Averaged Total score, used here, is calculated by averaging the three domain scores. Higher values represent a better outcome.
Time Frame: This outcome will be assessed via self-report instrument from the patient participant 6 months after discharge from inpatient rehabilitation care.
Population: Individuals with complete data for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan
Number analyzed (Participants) | 363 | 372
units on a scale | 1.30 (0.61) | 1.33 (0.57)
Statistical Analysis 1: Comparison: Rehabilitation Discharge Plan vs Rehabilitation Transition Plan; It was calculated that 500 to 900 participants randomized in a 1:1 fashion between the two arms would have practically 100% power to detect an effect size of 0.5, and even a small sample size of 300 would have 80% power to detect a small effect size of 0.3 (800 to 900 would be 100% power); Test type: Superiority; p = 0.44, t-test, 2 sided — The threshold for statistical significance was p = 0.05; t-test for independent samples, two-tailed, allocation ratio=1; Mean Difference (Net) = -0.78 — Intervention mean minus control mean

2. Primary Outcome: Quality of Life After Brain Injury Scale (QoLIBRI)
Description: A patient-reported instrument specifically created to measure the patient's perception of their health-related quality of life following TBI. The QOLIBRI scores are reported on a 0-100 scale, where 0=worst possible quality of life and 100=best possible quality of life.
Time Frame: as for outcome 1
Population: Participants with complete data for this measure. This measure could only be collected from the patient (no proxy data).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan
Number analyzed (Participants) | 291 | 315
score on a scale | 68.3 (19.3) | 65.9 (19.3)
Statistical Analysis 1: Comparison: Rehabilitation Discharge Plan vs Rehabilitation Transition Plan; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Net) = 1.63

3. Secondary Outcome: Cornell Services Index
Description: A patient-reported instrument created to assess healthcare services utilization. This reports the number and percentage of individuals who attended at least one visit of a specialty during follow-up, regardless of whether they had been recommended and/or scheduled at discharge.
Time Frame: This outcome will be assessed via self-report instrument from the patient participant 3, 6, 9 and 12 months after discharge from inpatient rehabilitation care.
Population: Individuals who had at least one follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan
Number analyzed (Participants) | 419 | 418
Participants
  Rehabilitation Medicine | 260 | 266
  Physical Therapy | 325 | 324
  Occupational Therapy | 262 | 283
  Primary Care Visits | 347 | 365
  Speech Therapy | 247 | 261
  Neurosurgery | 162 | 156
  Neuropsychology | 119 | 146
  Neurology: number analyzed (Participants) | 418 | 418
  Neurology | 210 | 217
  Neuro-optometry/Neuro-ophthalmology | 118 | 124
  Social Worker | 83 | 88
  Psychologist/Mental health | 104 | 120
  Vocational Counseling | 46 | 62
  Psychiatrist | 88 | 101
  Vision Therapy | 32 | 31

4. Secondary Outcome: Bakas Caregiving Outcomes Scale
Description: A 15-item measure, each with a 7-point scale that assesses change in social functioning, emotional well-being, and physical health related to caregiving. Item scores are transformed to 1-7, then summed to provide total scale scores ranging from 15 - 105, with a higher score indicating a better outcome.
Time Frame: This outcome was assessed via self-report instrument from the caregiver participant at 3, 6, 9 and 12 months after the patient is discharged from inpatient rehabilitation care. This is reporting the 6-month outcomes.
Population: Caregiver participants with complete data for the measure at the 6 month follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Number analyzed (Participants) | 225 | 228
score on a scale | 60.1 (15.1) | 60.0 (13.9)

5. Secondary Outcome: Zarit Burden Interview
Description: 12 item version addresses the concerns that our stakeholders feel are most important and that we feel are most relevant to our study interventions. The minimum and maximum values are 0 to 88, with 88 representing the most burden (worst outcome).
Time Frame: as for outcome 4
Population: Caregiver participants with complete data for the measure at the 6 month follow-up timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Number analyzed (Participants) | 223 | 233
units on a scale | 22.5 (15.3) | 22.8 (16.3)

6. Secondary Outcome: Short Form 12-Item Measure (SF-12)
Description: The SF-12 is a measure of health-related quality of life (HRQOL) and allows for 2 component scores to be determined: physical health and mental health. The scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Time Frame: as for outcome 4
Population: Caregiver participants with complete data for the measure at the 6 month follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Number analyzed (Participants) | 222 | 228
score on a scale
  Physical Component | 51.1 (10.0) | 50.1 (10.0)
  Mental Component | 46.0 (11.8) | 46.9 (11.7)

7. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Satisfaction With Social Roles and Activities 8a
Description: A measure that assesses engagement in roles and activities apart from those related to caregiving. Raw scores are converted to scale scores, with a range of 26.2 to 65.6, with the higher score indicating better outcome.
Time Frame: as for outcome 4
Population: Caregiver participants with complete data for the measure at the 6 month follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Number analyzed (Participants) | 228 | 234
score on a scale | 51.2 (9.0) | 50.3 (8.5)

8. Secondary Outcome: Time Spent Caregiving - Required Assistance
Description: A measure developed by the study team to describe the use of caregivers for individuals with TBI. The "Required Assistance" portion of the measure asks how much oversight or supervision the patient needs on a daily basis, ranging from 1) "Need someone in the room awake at all time" to 12) "Lives independently with minimal assistance". Responses were categorized into three levels with 1-8 equaling "Need supervision", 9-10 equaling "Need assistance", and 11-12 equaling "Independent".
Time Frame: as for outcome 4
Population: Caregiver participants with complete data for the measure at the 6 month follow-up timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Number analyzed (Participants) | 227 | 232
Participants
  Need supervision | 121 | 120
  Need assistance | 39 | 40
  Independent | 67 | 72

9. Secondary Outcome: Participation Assessment With Recombined Tools - Objective 17 (PART-O-17)
Description: as for outcome 1
Time Frame: This outcome will be assessed longitudinally via self-report instrument from the patient participant 3,6, 9 and 12 months after discharge from inpatient rehabilitation care.
Population: Total participants randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan
Number analyzed (Participants) | 462 | 463
score on a scale
  3 month: number analyzed (Participants) | 384 | 382
  3 month | 1.22 (0.56) | 1.20 (0.52)
  6 month: number analyzed (Participants) | 363 | 372
  6 month | 1.30 (0.61) | 1.33 (0.57)
  9 month: number analyzed (Participants) | 363 | 357
  9 month | 1.35 (0.60) | 1.34 (0.58)
  12 month: number analyzed (Participants) | 303 | 292
  12 month | 1.36 (0.61) | 1.35 (0.58)

10. Secondary Outcome: Quality of Life After Brain Injury Scale (QoLIBRI)
Description: as for outcome 2
Time Frame: as for outcome 3
Population: Total participants randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan
Number analyzed (Participants) | 462 | 463
score on a scale
  3 month: number analyzed (Participants) | 300 | 303
  3 month | 67.5 (18.1) | 65.1 (18.1)
  6 month: number analyzed (Participants) | 291 | 315
  6 month | 68.3 (18.1) | 65.9 (17.8)
  9 month: number analyzed (Participants) | 303 | 300
  9 month | 68.3 (19.9) | 66.0 (19.0)
  12 month: number analyzed (Participants) | 303 | 292
  12 month | 68.3 (20.2) | 65.8 (19.3)

11. Secondary Outcome: Satisfaction With Care
Description: A measure developed by the study team to assess satisfaction with health care received by the patient participant. Patients, caregivers, both, or another appropriate proxy could rate their satisfaction with different domain's of the patient's care on a 1-7 scale, where 1 = Very dissatisfied, 7 = Very satisfied, and 4 = Neutral. Higher scores indicate higher satisfaction (better outcome).
Time Frame: This outcome will be assessed via self-report instrument from the patient participant 6 and 12 months after discharge from inpatient rehabilitation care. 6-month outcomes are reported.
Population: Participants with complete data for this measure at 6 months post-discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan
Number analyzed (Participants) | 332 | 346
units on a scale
  Get help coordinating healthcare | 5.69 (1.71) | 5.74 (1.62)
  Attend appointments: number analyzed (Participants) | 332 | 345
  Attend appointments | 6.05 (1.45) | 5.99 (1.55)
  Get answers about healthcare: number analyzed (Participants) | 332 | 345
  Get answers about healthcare | 5.76 (1.59) | 5.81 (1.5)
  Connect with community resources/services: number analyzed (Participants) | 331 | 344
  Connect with community resources/services | 5.01 (1.83) | 5.27 (1.78)
  Receive help when it's needed | 5.72 (1.75) | 5.86 (1.62)

12. Secondary Outcome: RTP Satisfaction Survey
Description: A measure developed by the study team to assess satisfaction with RTP (intervention), measured through Likert-scaled and open-ended questions.
Time Frame: This outcome was assessed via self-report instrument from both patient and caregiver participants (if applicable) randomized to the RTP group 6 months after discharge from inpatient rehabilitation care (if they consented to complete the survey).
Population: The 16 patients and caregivers who jointly completed the survey are represented in both groups, however the data table shows data for the combined surveys only in the patient column, therefore the number of caregivers represented in the caregiver column is only 104.
Measure: Count of Participants; unit: Participants
Groups:
- RTP Survey - Patients: Patient participants who were eligible for and completed the RTP Satisfaction Survey. Of the 463 patient participants randomized to receive RTP, 154 were enrolled prior to the survey being added to the research protocol and were thus considered ineligible for the survey. In addition, 23 patient participants did not engage with the TCM and were therefore ineligible for the survey, and 26 patient participants withdrew from the study or expired. Out of 260 eligible, 175 (67%) completed the survey).
- RTP Survey - Caregivers: Caregiver participants who were eligible for and completed the RTP Satisfaction Survey. Of the 295 caregiver participants randomized to receive RTP, 100 caregivers were enrolled prior to the survey being added to the research protocol and were thus considered ineligible for the survey. In addition, 21 caregiver participants did not engage with the TCM and were therefore ineligible for the survey, and 18 caregiver participants withdrew from the study or expired. Out of 157 eligible, 120 (76%) completed the survey.
Arm/Group | RTP Survey - Patients | RTP Survey - Caregivers
Number analyzed (Participants) | 175 | 120
Participants
  RTP helped with resources connections after discharge: number analyzed (Participants) | 175 | 104
  RTP helped with resources connections after discharge: Not at all | 5 | 3
  RTP helped with resources connections after discharge: A little bit | 14 | 5
  RTP helped with resources connections after discharge: Moderately | 29 | 13
  RTP helped with resources connections after discharge: A lot | 40 | 24
  RTP helped with resources connections after discharge: Extremely | 68 | 57
  RTP helped with resources connections after discharge: NA/Not Answered | 19 | 2
  RTP helped with practical, day-to-day adjustment to life with a brain injury: number analyzed (Participants) | 175 | 104
  RTP helped with practical, day-to-day adjustment to life with a brain injury: Not at all | 6 | 3
  RTP helped with practical, day-to-day adjustment to life with a brain injury: A little bit | 13 | 5
  RTP helped with practical, day-to-day adjustment to life with a brain injury: Moderately | 33 | 15
  RTP helped with practical, day-to-day adjustment to life with a brain injury: A lot | 57 | 23
  RTP helped with practical, day-to-day adjustment to life with a brain injury: Extremely | 54 | 52
  RTP helped with practical, day-to-day adjustment to life with a brain injury: NA/Not Answered | 12 | 6
  RTP helped with emotional adjustment to life with a brain injury: number analyzed (Participants) | 175 | 104
  RTP helped with emotional adjustment to life with a brain injury: Not at all | 12 | 4
  RTP helped with emotional adjustment to life with a brain injury: A little bit | 12 | 3
  RTP helped with emotional adjustment to life with a brain injury: Moderately | 33 | 11
  RTP helped with emotional adjustment to life with a brain injury: A lot | 44 | 29
  RTP helped with emotional adjustment to life with a brain injury: Extremely | 63 | 54
  RTP helped with emotional adjustment to life with a brain injury: NA/Not Answered | 11 | 3
  RTP helped accomplish the things you wanted to do: number analyzed (Participants) | 175 | 104
  RTP helped accomplish the things you wanted to do: Not at all | 8 | 4
  RTP helped accomplish the things you wanted to do: A little bit | 14 | 7
  RTP helped accomplish the things you wanted to do: Moderately | 30 | 21
  RTP helped accomplish the things you wanted to do: A lot | 51 | 25
  RTP helped accomplish the things you wanted to do: Extremely | 53 | 42
  RTP helped accomplish the things you wanted to do: NA/Not Answered | 19 | 5
  It was valuable to talk with someone who understands TBI: number analyzed (Participants) | 175 | 104
  It was valuable to talk with someone who understands TBI: Not at all | 3 | 3
  It was valuable to talk with someone who understands TBI: A little bit | 4 | 0
  It was valuable to talk with someone who understands TBI: Moderately | 10 | 3
  It was valuable to talk with someone who understands TBI: A lot | 30 | 12
  It was valuable to talk with someone who understands TBI: Extremely | 120 | 83
  It was valuable to talk with someone who understands TBI: NA/Not Answered | 8 | 3

13. Secondary Outcome: Time Spent Caregiving - Reason for Assistance
Description: The "Reason for Assistance" measure asks which category captures the reason the patient cannot be alone (if in the "Need supervision" or "Need assistance" category for Required Assistance).
Time Frame: as for outcome 4
Population: Caregivers who reported the patient in the "Need supervision" or "Need assistance" category for Required Assistance measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers
Number analyzed (Participants) | 159 | 161
Participants
  Cognition/Behavior | 39 | 42
  Physical function | 33 | 32
  Both | 82 | 83
  Other | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the participant's participation, approximately 12 months.
Description: Adverse events were recorded when brought up by participants during data collection and intervention activities, and categorized as Serious or non-serious. SAE's were categorized into five categories: Death, life threatening, hospitalization - initial or prolonged, disability/incapacity, or required intervention to prevent permanent impairment. Each event had a brief description of the nature collected. No events were determined to be related to study activities.
Groups:
- Death Prior to Randomization: Patient who expired after enrollment but prior to randomization.
Arm/Group | Rehabilitation Discharge Plan | Rehabilitation Transition Plan | Rehabilitation Discharge Plan - Caregivers | Rehabilitation Transition Plan - Caregivers | Death Prior to Randomization
All-Cause Mortality (participants affected / at risk) | 14/462 | 21/463 | 3/296 | 1/295 | 1/11
Serious Adverse Events (participants affected / at risk) | 127/462 | 141/463 | 4/296 | 9/295 | 0/11
Other Adverse Events (participants affected / at risk) | 107/462 | 158/463 | 10/296 | 13/295 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rehabilitation Discharge Plan (N=462) | Rehabilitation Transition Plan (N=463) | Rehabilitation Discharge Plan - Caregivers (N=296) | Rehabilitation Transition Plan - Caregivers (N=295) | Death Prior to Randomization (N=11)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Cardiac disorders (Cardiac disorders) | 3 (3) | 12 (16) | 0 (0) | 0 (0) | NA
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (8) | 4 (4) | 0 (0) | 0 (0) | NA
General disorders (General disorders) | 25 (25) | 27 (31) | 2 (2) | 3 (3) | NA — Events that do not fall into a specific category
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | NA
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Infections and infestations (Infections and infestations) | 30 (37) | 25 (31) | 0 (0) | 1 (1) | NA
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 24 (29) | 20 (20) | 0 (0) | 1 (1) | NA
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 (7) | 5 (5) | 0 (0) | 1 (1) | NA
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (5) | 0 (0) | 1 (1) | NA
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Nervous system disorders (Nervous system disorders) | 35 (53) | 48 (71) | 0 (0) | 0 (0) | NA
Psychiatric disorders (Psychiatric disorders) | 11 (12) | 17 (18) | 0 (0) | 0 (0) | NA
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | NA
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 9 (11) | 0 (0) | 0 (0) | NA
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | NA
Surgical and medical procedures (Surgical and medical procedures) | 8 (9) | 9 (10) | 0 (0) | 0 (0) | NA
Vascular disorders (Vascular disorders) | 6 (6) | 9 (13) | 1 (1) | 2 (2) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rehabilitation Discharge Plan (N=462) | Rehabilitation Transition Plan (N=463) | Rehabilitation Discharge Plan - Caregivers (N=296) | Rehabilitation Transition Plan - Caregivers (N=295) | Death Prior to Randomization (N=11)
Cardiac disorders (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | NA
Endocrine disorders (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Eye disorders (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | NA
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (7) | 13 (14) | 1 (1) | 0 (0) | NA
General disorders (General disorders) | 5 (5) | 12 (14) | 0 (0) | 0 (0) | NA
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | NA
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Infections and infestations (Infections and infestations) | 21 (23) | 28 (32) | 5 (5) | 7 (7) | NA
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 42 (46) | 54 (65) | 2 (2) | 3 (3) | NA
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | NA
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 7 (8) | 12 (15) | 1 (1) | 1 (1) | NA
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | NA
Nervous system disorders (Nervous system disorders) | 16 (18) | 21 (24) | 0 (0) | 0 (0) | NA
Psychiatric disorders (Psychiatric disorders) | 5 (7) | 7 (9) | 1 (1) | 0 (0) | NA
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | NA
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 0 (0) | 0 (0) | NA
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | NA
Surgical and medical procedures (Surgical and medical procedures) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | NA
Vascular disorders (Vascular disorders) | 4 (4) | 8 (8) | 0 (0) | 0 (0) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03422276/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Consent (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03422276/ICF_001.pdf
  • Informed Consent Form: Caregiver Consent (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03422276/ICF_002.pdf